CLINICAL TRIAL: NCT03627260
Title: How Useful is the Advice: "Fill up a Handful of Sunscreen and Spread it All Over Your Body"
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bispebjerg Hospital (Other)
Responsible Party: Principal Investigator, Ida M. Heerfordt, Principal Investigator, Bispebjerg Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: Handful of sunscreen
Record Dates: First submitted 2018-03-07; First posted 2018-08-13 (Actual); Last update posted 2018-08-13 (Actual); Status verified 2018-08

CONDITIONS: Quantity of Sunscreen; Sun Protection Factor; Sun Safety Campaigns; Sunscreen Use

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Behavioral: Fill up a handful of sunscreen and spread it all over your body. Sunscreen, Actinica — Volunteers were asked to follow the rule of thumb: "Fill up a handful of sunscreen and spread it all over your body".

SUMMARY:
The advice: "Fill up a handful of sunscreen and spread it all over your body" is used in several sun safety campaigns. The hope is that users in swimwear following the advice will apply a sunscreen quantity of 2 mg/cm^2 to all accessible skin. The present study is the first to investigate how this advice works in practice.

ELIGIBILITY:
Inclusion Criteria:

- European descent

Exclusion Criteria:

* Skin disease
* allergy to the content in sunscreen
* Pregnancy
* Breastfeeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2017-05-01 (Actual); Primary Completion 2017-07-29 (Actual); Study Completion 2017-07-29 (Actual)

PRIMARY OUTCOMES:
The overall quantities of sunscreen applied were calculated from the weighed amount of sunscreen used divided by the skin area accessible for sunscreen application. | Outcome measure will be assessed within half an hour after sunscreen application. There will be no further follow up.

CONTACTS AND LOCATIONS:
Locations (1):
- Bispebjerg Hospital, Copenhagen NV, DK, Denmark